CLINICAL TRIAL: NCT06168981
Title: The Effect of Preoperative Chewing Gum on Anxiety and Sore Throat in Patients With Laryngeal Mask Airway: A Randomised Controlled Trial
Brief Title: The Effect of Preoperative Chewing Gum on Anxiety and Sore Throat in Patients With Laryngeal Mask Airway
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Neslihan Ilkaz, Assistant Professor, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023/197
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Laryngeal Mask; Throat Pain; Anxiety
Keywords: Laryngeal mask; Pain; Chewing gum; Anxiety
MeSH Terms: conditions — Pharyngitis; Anxiety Disorders; Pain | interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chewing Gum (Experimental): Before the surgery, the patient will chew gum for 2 minutes and routine nursing care will be applied. Anxiety level will be evaluated before and after chewing gum.
  Interventions: Other: Chewing Gum
- Control Group (No Intervention): Anxiety level will be evaluated before and after routine nursing care.

INTERVENTIONS:
Other: Chewing Gum — The patient will be asked to chew gum before the surgery during the 2 minutes. Anxiety level will evaluated before and after chewing gum.
  Arms: Chewing Gum

SUMMARY:
This study was planned to investigate the effect of chewing gum in the preoperative period on patients' sore throat and anxiety levels.

DETAILED DESCRIPTION:
Postoperative sore throat is a common complaint (1,2). It is reported in the literature that there are various pharmacological methods to reduce this condition, such as the use of nebula, corticosteroids, nonsteroidal anti-inflammatory drugs, or lidocaine. However, these methods have various advantages and disadvantages (3,4). Chewing gum, one of the non-pharmacological methods may be safer for the patient. Chewing gum increases salivary gland secretion and provides lubrication of the oral cavity (5). For this reason, it was thought that chewing gum before surgery could reduce throat pain after using a laryngeal mask due to the effect it provides. It has been determined that there are few experimental studies on the subject in the literature (6,7).

The presence of preoperative anxiety may lead to an increase in the need for intraoperative anesthesia and analgesic consumption in the postoperative period (8,9). However, it may cause a decrease in patient satisfaction and prolong the recovery process in the postoperative period (8,9). Pharmacological approaches can be applied to address this concern. However, non-pharmacological approaches may be safer for patients. Chewing gum during this process can also reduce patients' anxiety levels. A sufficient number of studies on the subject could not be found (10).

The study will conduct as a prospective randomized controlled trial. After obtaining verbal and written consent from the patients before and after the surgery, the study will conduct with various data collection forms.

These forms are; patient Identification form, Amsterdam Preoperative Anxiety and Information Scale (APAIS), Visual Analogue Scale (VAS). Patients will randomize. The chewing gum group in group- I (n=46), and group II (n=46) will be the control group. We have two stage.In first stage; anxiety levels will be measured for both group. In second stage; throat pain will evaluated at 2.-4.-6. hours.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective surgery
* Being intubated with a laryngeal mask
* Being ASA (American Society of Anesthesiologists) I-II

Exclusion Criteria:

* Using cigarette

  * Having asthma
  * Having chronic laryngitis
  * Having gastroesophageal reflux
  * Steroid use in the preoperative or intraoperative period
  * Mallampati score greater than two

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients will undergo breast surgery
Enrollment: 92 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from preoperative anxiety level in a 2 minutes | After chewing gum for 2 minutes
  In this section, the anxiety level will decrease or disappear. This status will evaluate with Amsterdam Preoperative Anxiety and Information Scale (APAIS). APAIS consists of two scales, including a four-item anxiety scale and two-items information requirement. Items are rated on a Likert scale from 1 ("not at all worried") to 5 ("very worried"). The score ranges for the anxiety subscale and the information need subscale are 4-20 and 2-10, respectively. High scores are associated with higher levels of anxiety and need for information. Cronbach's α coefficients for the anxiety subscale and the information need subscale were 0.86 and 0.68, respectively (Moerman et al.1996).
  Çetinkaya et al. The validity and reliability of the Turkish translation of APAIS was verified in 2019. Cronbach's α coefficients of the APAIS anxiety and information need subscales were 0.897 and 0.786, respectively

SECONDARY OUTCOMES:
Change from postoperative throat pain level at 2., 4., 6. hours | Time frame: Postoperative time at 2., 4., 6., hours
  In this section, the degree of postoperative throat pain level will decrease or disappear. This status will evaluate with Visual Analogue Scale (VAS). VAS is a horizontal line with a length of 10 cm. According to VAS, 0 is the lowest level and 10 is the highest level.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Ilkaz, PhD, Principal Investigator — Ankara Medipol University
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Medipol University, Ankara, Keçiören
  - Neslihan Ilkaz, Ankara, Keçiören

REFERENCES:
- [Background] Segaran S, Bacthavasalame AT, Venkatesh RR, Zachariah M, George SK, Kandasamy R. Comparison of Nebulized Ketamine with Nebulized Magnesium Sulfate on the Incidence of Postoperative Sore Throat. Anesth Essays Res. 2018 Oct-Dec;12(4):885-890. doi: 10.4103/aer.AER_148_18. PMID 30662125
- [Background] Miller DM, Camporota L. Advantages of ProSeal and SLIPA airways over tracheal tubes for gynecological laparoscopies. Can J Anaesth. 2006 Feb;53(2):188-93. doi: 10.1007/BF03021826. PMID 16434761
- [Background] Yu J, Ren L, Min S, Yang Y, Lv F. Nebulized pharmacological agents for preventing postoperative sore throat: A systematic review and network meta-analysis. PLoS One. 2020 Aug 10;15(8):e0237174. doi: 10.1371/journal.pone.0237174. eCollection 2020. PMID 32776966
- [Background] Wang G, Qi Y, Wu L, Jiang G. Comparative Efficacy of 6 Topical Pharmacological Agents for Preventive Interventions of Postoperative Sore Throat After Tracheal Intubation: A Systematic Review and Network Meta-analysis. Anesth Analg. 2021 Jul 1;133(1):58-67. doi: 10.1213/ANE.0000000000005521. PMID 33886521
- [Background] Hashiba T, Takeuchi K, Shimazaki Y, Takeshita T, Yamashita Y. Chewing xylitol gum improves self-rated and objective indicators of oral health status under conditions interrupting regular oral hygiene. Tohoku J Exp Med. 2015 Jan;235(1):39-46. doi: 10.1620/tjem.235.39. PMID 25744362
- [Background] 6. Abdelgalil, A. S., Abdelrahman, A. S., & Hassan, M. E. (2023). Preoperative gum chewing for different durations to prevent postoperative sore throat after endotracheal intubation: A randomized controlled trial. Trends in Anaesthesia and Critical Care, 101216.
- [Background] Zemla AJ, Nowicka-Sauer K, Jarmoszewicz K, Wera K, Batkiewicz S, Pietrzykowska M. Measures of preoperative anxiety. Anaesthesiol Intensive Ther. 2019;51(1):64-69. doi: 10.5603/AIT.2019.0013. PMID 31280554
- [Background] Stamenkovic DM, Rancic NK, Latas MB, Neskovic V, Rondovic GM, Wu JD, Cattano D. Preoperative anxiety and implications on postoperative recovery: what can we do to change our history. Minerva Anestesiol. 2018 Nov;84(11):1307-1317. doi: 10.23736/S0375-9393.18.12520-X. Epub 2018 Apr 5. PMID 29624026
- [Background] Bang YJ, Lee JH, Kim CS, Lee YY, Min JJ. Anxiolytic effects of chewing gum during preoperative fasting and patient-centered outcome in female patients undergoing elective gynecologic surgery: randomized controlled study. Sci Rep. 2022 Mar 9;12(1):4165. doi: 10.1038/s41598-022-07942-6. PMID 35264684